CLINICAL TRIAL: NCT05815719
Title: Continuous Ovarian Stimulation in DUOSTIM Cycles.
Brief Title: Continuous Double Ovarian Stimulation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Juan Carlos Castillo, Principal investigator, Instituto Bernabeu
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBMR31; 2022-003177-32 (EudraCT Number)
Record Dates: First submitted 2023-03-23; First posted 2023-04-18 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Fertility Issues
Keywords: OVARIAN STIMULATION
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin alfa; Urofollitropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients to carry out an experimental double ovarian stimulation and to receive 4 weekly injections of Corifollitropin alfa. Prospective group.
  Interventions: Drug: Corifollitropin Alfa
- Control group (Active Comparator): Patients to carry out a conventional double ovarian stimulation and to receive daily injections of gonadotropins. Retrospective group (data retrieved from strictly selected treatments carried out in our institution within the 24 months prior to the inclusion of the first patient in the study group and according to the standard guideline of the clinic).
  Interventions: Drug: Follitropin Alfa; Drug: Follitropin Alfa Biosimilar; Drug: Urinary Human follicle stimulating hormone

INTERVENTIONS:
Drug: Corifollitropin Alfa — 150 micrograms per dose
  Other Names: 4 Weekly Corifollitropin Alfa injections
  Arms: Study group
Drug: Follitropin Alfa — Variable dose.
  Other Names: Daily injections of gonadotropins
  Arms: Control group
Drug: Follitropin Alfa Biosimilar — Variable dose.
  Other Names: Daily injections of gonadotropins
  Arms: Control group
Drug: Urinary Human follicle stimulating hormone — Variable dose.
  Other Names: Daily injections of gonadotropins
  Arms: Control group

SUMMARY:
To evaluate the efficacy of the weekly use of corifollitropin alfa in double ovarian stimulation process and to compare it to the conventional protocol with daily medication administration.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the efficacy of the weekly use of corifollitropin alfa in terms of ovarian stimulation results and its biological outcomes (total number of oocytes retrieved) in case of ovarian stimulation cycles in double stimulation modality (DUOSTIM) and in comparison with the conventional DUOSTIM protocol: daily administration of gonadotropins.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for DUOSTIM protocol
* Maximum age of 43 years (up to one day before their 44th birthday) at the beginning of the stimulation process.
* Ability to participate and comply with the study protocol.
* To have given written consent

Exclusion Criteria:

* Finding of ovarian pathology at the time of initiation of stimulation: e.g. ovarian cysts.
* Concurrent participation in another study.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Given the aim is to carry out ovarian stimulation, only persons with female reproductive system can be eligible.
Enrollment: 30 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Castillo Farfan, MD, PhD, Principal Investigator — Instituto Bernabeu
Locations (1):
- Instituto Bernabeu, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
The PI will collect individual data which will later be analyzed. Only analyzed overall data will be shared.

REFERENCES:
- [Result] Baerwald AR, Adams GP, Pierson RA. Characterization of ovarian follicular wave dynamics in women. Biol Reprod. 2003 Sep;69(3):1023-31. doi: 10.1095/biolreprod.103.017772. Epub 2003 May 14. PMID 12748128
- [Result] Devroey P, Boostanfar R, Koper NP, Mannaerts BM, Ijzerman-Boon PC, Fauser BC; ENGAGE Investigators. A double-blind, non-inferiority RCT comparing corifollitropin alfa and recombinant FSH during the first seven days of ovarian stimulation using a GnRH antagonist protocol. Hum Reprod. 2009 Dec;24(12):3063-72. doi: 10.1093/humrep/dep291. Epub 2009 Aug 14. PMID 19684043
- [Result] Kuang Y, Chen Q, Hong Q, Lyu Q, Ai A, Fu Y, Shoham Z. Double stimulations during the follicular and luteal phases of poor responders in IVF/ICSI programmes (Shanghai protocol). Reprod Biomed Online. 2014 Dec;29(6):684-91. doi: 10.1016/j.rbmo.2014.08.009. Epub 2014 Sep 6. PMID 25444501
- [Result] Kuang Y, Hong Q, Chen Q, Lyu Q, Ai A, Fu Y, Shoham Z. Luteal-phase ovarian stimulation is feasible for producing competent oocytes in women undergoing in vitro fertilization/intracytoplasmic sperm injection treatment, with optimal pregnancy outcomes in frozen-thawed embryo transfer cycles. Fertil Steril. 2014 Jan;101(1):105-11. doi: 10.1016/j.fertnstert.2013.09.007. Epub 2013 Oct 23. PMID 24161646
- [Result] Vaiarelli A, Cimadomo D, Petriglia C, Conforti A, Alviggi C, Ubaldi N, Ledda S, Ferrero S, Rienzi L, Ubaldi FM. DuoStim - a reproducible strategy to obtain more oocytes and competent embryos in a short time-frame aimed at fertility preservation and IVF purposes. A systematic review. Ups J Med Sci. 2020 May;125(2):121-130. doi: 10.1080/03009734.2020.1734694. Epub 2020 Apr 25. PMID 32338123
- [Result] Vaiarelli A, Cimadomo D, Trabucco E, Vallefuoco R, Buffo L, Dusi L, Fiorini F, Barnocchi N, Bulletti FM, Rienzi L, Ubaldi FM. Double Stimulation in the Same Ovarian Cycle (DuoStim) to Maximize the Number of Oocytes Retrieved From Poor Prognosis Patients: A Multicenter Experience and SWOT Analysis. Front Endocrinol (Lausanne). 2018 Jun 14;9:317. doi: 10.3389/fendo.2018.00317. eCollection 2018. PMID 29963011
- [Derived] Castillo JC, Fuentes A, Ortiz JA, Abellan E, Bernabeu A, Bernabeu R. Continuous ovarian stimulation: a proof-of-concept study exploring the uninterrupted use of corifollitropin alpha in DuoStim cycles for enhanced efficiency and patient convenience (Alicante protocol). F S Rep. 2024 Mar 28;5(2):176-182. doi: 10.1016/j.xfre.2024.03.005. eCollection 2024 Jun. PMID 38983736

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled patients all had to comply with the entry criteria and were all assiged to the "study group". The "control group" subjects were selected restrospectively by also complying with the criteria and with similar characteristics (such as AMH level, BMI, age) to the "study group" ones.
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Retrieved Oocytes
Description: To investigate the total number of oocytes retrieved through ovarian stimulation in double ovarian stimulation cycles (DUOSTIM) utilizing weekly subcutaneous injections of Corifollitropin alfa (study group) vs. daily injections of gonadotropins (control group).
Time Frame: Through study completion, an average of four weeks
Measure: Mean (Standard Deviation); unit: oocytes
Groups:
- Control Group: Patients that have carried out standard double ovarian stimulation and received daily injections of gonadotropins. Retropective group.
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 15 | 15
oocytes | 13.33 (6.904) | 11.87 (6.105)

2. Primary Outcome: Number of MII Oocytes
Description: To compare the total number of MII oocytes obtained in double stimulation cycles in study vs control groups
Time Frame: Through study completion, an average of four months
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 15 | 15
oocytes | 10.4 (6.3) | 9.2 (4.6)

3. Secondary Outcome: Duration of Ovarian Stimulation
Description: Total days of follicular and luteal phases
Time Frame: Through study completion, an average of four months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 15 | 15
days | 24.4 (3.5) | 25.2 (4.9)

4. Secondary Outcome: Number of Injections
Description: Number of injections during the DUOSTIM cycle
Time Frame: Through study completion, an average of four months
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 15 | 15
injections | 4.5 (1.4) | 35.2 (12.2)

ADVERSE EVENTS:
Time Frame: 45 days. From the start of ovarian stimulation to one week after the second oocyte retrieval in the DUOSTIM cycle.
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
The limitations of the present study correspond to the comparative with historical records and not blinding the patients. in addition, the study does not evaluate data on oocyte quality beyond fertilization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT05815719/Prot_SAP_000.pdf